CLINICAL TRIAL: NCT05605171
Title: Impact of Posterior Urethrovesical Reconstruction on Early Return to Urinary Continence Following Robot-assisted Radical Prostatectomy: a Prospective Randomized Controlled Trial
Brief Title: Posterior Urethrovesical Anastomotic Reconstruction in Comparison to Conventional Urethrovesical Anastomosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Bobby Shayegan, Associate Professor & Head, David Braley & Nancy Gordon Chair in Urology, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BFCRS-RP-U-01a
Record Dates: First submitted 2022-10-23; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer
Keywords: Localized prostate cancer; Robot-assisted laparoscopic radical prostatectomy; Vesicourethral anastomosis; Posterior vesicourethral anastomosis reconstruction; Rocco stitch; Urinary incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior reconstruction urethrovesical anastomosis. (Experimental): The intervention comprised of a 2-stitch approximation of the free edge of the Denonvilliers' fascia and posterior bladder wall cranially, to the posterior aspect of the rhabdosphincter and the posterior median raphe caudally, respectively, following prostate extraction. The aim of this approach is to ultimately restore the length of the urethrosphincteric complex, prevent its caudal retraction, and avoid undue tension on the subsequent vesicourethral anastomosis, and provide a posterior support to the urethral sphincter complex to facilitate its effective contraction.
  Interventions: Procedure: Posterior reconstruction urethrovesical anastomosis.
- Conventional urethrovesical anastomosis. (Active Comparator): The conventional is fashioned with a continuous running technique that uses two sutures. The first suture is passed in a clockwise hemicircumferential manner, starting from outside in on the bladder neck at the 5 o'clock position and inside out on the urethra up toward the 12 o'clock position. The second suture is similarly run in a counter- clockwise hemicircumferential direction. The running sutures are snug down after each apposition to ensure there is no slack, and finally tied together with several knots at the 12 o'clock position.
  Interventions: Procedure: Conventional vesicourethral anastomosis.

INTERVENTIONS:
Procedure: Posterior reconstruction urethrovesical anastomosis. — Rocco stitch.
  Arms: Posterior reconstruction urethrovesical anastomosis.
Procedure: Conventional vesicourethral anastomosis. — Standard of care.
  Arms: Conventional urethrovesical anastomosis.

SUMMARY:
Urinary incontinence post radical prostatectomy is a well-recognized complication regardless of approach, with a potential negative impact on health-related quality of life. Although 12-month continence rates range from 85-95% in the literature, few patients are continent in the early postoperative period. It has been suggested that posterior reconstruction of the Denonvilliers' musculofascial plate, also known as the Rocco stitch, may improve early return to urinary continence, though clinical equipoise remains.

DETAILED DESCRIPTION:
Each modality of prostate cancer treatment has the propensity to lead to negative outcomes on quality of life to varying degrees. It is our responsibility to incorporate into our practices the most beneficial treatment regimens that render patients' cancer-free while minimizing potential treatment-related adverse outcomes, including incontinence and erectile dysfunction. Urinary incontinence and erectile dysfunction are the two most well described complications of radical prostatectomy with observed rates of 8.4% and 59.9%, respectively. Delayed recovery of urinary continence following radical prostatectomy (RP) is a well-known entity. Numerous contributing factors have been identified for post-prostatectomy incontinence (PPI), including both patient (age, body mass index, membranous urethral length, prostate volume, pre-existing lower urinary tract symptoms, and oncologic factors) and surgeon characteristics (experience, technique).

In a systematic review a meta-analysis using a no pad or a single safety pad definition, Ficcara and colleagues showed that the 12-month urinary incontinence rates can range from 8% to 11%. As such, several reconstructive options have been incorporated into the contemporary RP to attempt to improve these outcomes. The anatomy of urethral-sphincteric vesico-prostatic complex is well-described, leading to attempts to perform reconstruction of the Denonvilliers' musculofascial plate during the urethrovesical anastomosis (UVA) at the time of RP. Performing a posterior reconstruction (PR) of the rhabdosphincter was first reported by Rocco et al. in 2006 during open retropubic RP, showing a 3, 30, and 90-day improvement in urinary continence post catheter removal.

Posterior reconstruction urethrovesical anastomosis (PR-UVA) has been hypothesized to improve the integrity of the rhabdosphincter and potentially increase the functional urethral length. However, a recent systematic review evaluating the efficacy of PR-UVA showed no improvement in urinary continence at 1 week and 3, 6, and 12 months. Conflicting studies within the literature render an environment of clinical equipoise in this specific patient-related outcome. Our study objective was to address the true clinical benefit of the PR-UVA in a large prospective randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Any patient over age 18 (with the ability to give informed consent) with localized prostate cancer (cT1-2, N0, M0).

Exclusion Criteria:

* History of previous prostatic and/or urethral surgery
* A known history of a disease or comorbidity that could affect continence, such as insulin-dependent diabetes or urethral stenosis
* Presence of a urinary catheter preventing preoperative evaluation of continence.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2019-03-23 (Actual)

PRIMARY OUTCOMES:
Return to urinary incontinence | 12 months post procedure
  The validated EPIC-26 (The Expanded Prostate Cancer Index Composite) Short Form (© The University of Michigan).

SECONDARY OUTCOMES:
Need for incontinence improving procedure | 5 years post surgery
  Midurethral sling or artificial urinary sphincter

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Shayegan, MD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No